CLINICAL TRIAL: NCT07233083
Title: External Oblique Intercostal Plane Block for Postoperative Analgesia in Liver Transplantation
Brief Title: External Oblique Intercostal Plane Block for Liver Transplantation Recipient
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: anestezi 5
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Liver Transplantation; Recipients of Liver Transplant; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External oblique intercostal plane block group (Active Comparator): The patients in the External Oblique Intercostal Plane Block group will receive bilateral external oblique intercostal plane block and patient controlled analgesia (PCA) with morphine for postoperative analgesia.
  Interventions: Other: External Oblique Intercostal Plane Block
- Control Group (Sham Comparator): The patients in the Control group will not receive any regional block and will receive patient controlled analgesia (PCA) with morphine for postoperative analgesia.
  Interventions: Other: Sham Procedure

INTERVENTIONS:
Other: External Oblique Intercostal Plane Block — External oblique intercostal plane block will be administered at the end of the surgery and after skin closure
  Arms: External oblique intercostal plane block group
Other: Sham Procedure — Sham Block (Ultrasound probe placement without needle insertion or injection)
  Arms: Control Group

SUMMARY:
Postoperative pain management is one of the key factors in improving rehabilitation and accelerating recovery. The external oblique intercostal plane block can be used to provide abdominal wall analgesia for effective pain control in abdominal surgery.

The aim of this study is to investigate the postoperative analgesic efficacy of the external oblique intercostal plane block in liver transplant recipients.

The investigators will compare a group receiving the external oblique intercostal plane block with a control group to determine whether this block provides effective postoperative analgesia in liver transplant recipients.

DETAILED DESCRIPTION:
Patients scheduled for liver transplantation will be separated into 2 groups: External Oblique Intercostal Plane Block Group and Control Group.

Patients in the External Oblique Intercostal Plane Block Group will be performed bilateral External Oblique Intercostal Plane Block at the end of the surgery and after skin closure and will receive patient controlled analgesia with morphine for postoperative analgesia.

Patients in the Control Group will not receive any block procedure and will receive patient controlled analgesia with morphine for postoperative analgesia.

Morphine consumption for first postoperative 48 hours, visual analog scale scores, time to need for first rescue analgesia, amount of rescue analgesic drug, incidence of postoperative nausea and vomiting, and Quality of Recovery-15 scores will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 to 75 years
* Scheduled for elective orthotopic liver transplantation (living or deceased donor)
* J-shaped or Mercedes incision planned
* ASA physical status III-IV
* Normal or acceptable coagulation profile at the time of block application (INR ≤ 1.5, platelet count ≥ 50,000/mm³, fibrinogen ≥ 150 mg/dL)
* Able to provide written informed consent

Exclusion Criteria:

* Coagulopathy at the time of block application (INR > 1.5, platelet count < 50,000/mm³, or fibrinogen < 150 mg/dL)
* Known allergy or hypersensitivity to local anesthetics (amide group)
* Local infection or skin lesion at the block injection site
* Severe hemodynamic instability requiring high-dose vasopressor support
* Chronic opioid use (≥30 mg oral morphine equivalents per day for ≥30 days before surgery)
* Severe hepatic encephalopathy or cognitive impairment preventing use of PCA or pain scoring
* Emergency or re-transplantation surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The amount of morphine required by the patient and given by the device will be recorded for the first 24 hours | Postoperative 24 hours

SECONDARY OUTCOMES:
Postoperative visual analog scale scores | Postoperative 24 hours
  Postoperative pain will be assessed using a visual analog scale (VAS) (from 0 = no pain to 10 = maximum possible pain) for the first 24 hours.
Rescue analgesic drug consumption | postoperative 24 hours
  The amount of rescue analgesic in mg required by the patient will be recorded for the first 24 hours
Incidence of postoperative nausea and vomiting | postoperative 24 hours
  Number of patients developing postoperative nausea and vomiting will be recorded for the first 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided